CLINICAL TRIAL: NCT00970294
Title: Feasibility and Effectiveness of a Health Promotion Program on Aerobic Fitness and Glycemic Control for Adults With Type 2 Diabetes
Brief Title: Pilot Project of Health Promotion for People With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patricia Kluding, PhD (Other)
Responsible Party: Sponsor-Investigator, Patricia Kluding, PhD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 10946
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health Promotion Program (Experimental): Supervised exercise, educational sessions, dietary counseling
  Interventions: Behavioral: Health Promotion Program

INTERVENTIONS:
Behavioral: Health Promotion Program — 10 week health promotion program 3-4 times per week

SUMMARY:
Limited participation in health promotion activities is noted in people with diabetes, even though lifestyle changes have been found to be essential in decreasing the risk of complications of the disease. The purpose of this study is to gather preliminary data to assess the feasibility of an intense, customized health promotion program in people with diabetes, and to evaluate outcome measures following participation to determine effect size for future studies. Subjects with type 2 diabetes will participate in a 10-week health promotion program, at a frequency of 3-4 days per week. The intervention will include aerobic and strength training exercises with a schedule of progression, individual nutrition counseling, and diabetes health education sessions.

ELIGIBILITY:
Inclusion Criteria:

1. diabetes type II
2. age 40-70

Exclusion Criteria:

1. hospitalization for myocardial infarction, heart surgery, or congestive heart failure during the preceding 3 months
2. significant cardiac arrythmia, hypertrophic cardiomyopathy, severe aortic stenosis, or pulmonary embolus
3. recent symptoms of chest discomfort
4. currently smoking or significant pulmonary pathology
5. serious musculoskeletal problems that would limit ability to exercise
6. current active involvement in a regular exercise program (> 3 times per week)
7. open wounds on the weight bearing surface of the feet
8. not able to ambulate independently
9. stroke or other central nervous system pathology
10. stage 2 hypertension (resting blood pressure > 160 systolic or > 100 diastolic)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kluding, PhD, Study Director — University of Kansas Medical Center
Locations (1):
- Patricia Kluding PhD, Kansas City, Kansas, United States

REFERENCES:
- [Result] Kluding PM, Singh R, Goetz J, Rucker J, Bracciano S, Curry N. Feasibility and effectiveness of a pilot health promotion program for adults with type 2 diabetes: lessons learned. Diabetes Educ. 2010 Jul-Aug;36(4):595-602. doi: 10.1177/0145721710370718. Epub 2010 Jun 8. PMID 20530663

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health Promotion Program
Started | 11
Completed | 6
Not Completed | 5
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Health Promotion Program
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 58.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Recruitment, Retention, Adherence
Description: % of enrolled subjects who completed the trial
Time Frame: 10 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Health Promotion Program
Number analyzed (Participants) | 11
percentage of participants | 55

2. Secondary Outcome: Aerobic Fitness
Description: peak VO2 as measured with a graded maximal exercise test on a cycle ergometer
Time Frame: Baseline and at 10 weeks (change score)
Measure: Mean (Standard Deviation); unit: mL/kg/m
Arm/Group | Health Promotion Program
Number analyzed (Participants) | 6
mL/kg/m | 0.75 (1.78)

3. Secondary Outcome: Glycemic Control
Description: HbA1c measure
Time Frame: Baseline and at 10 weeks (change score)
Measure: Mean (Standard Deviation); unit: percentage of glycosolated hemoglobin
Arm/Group | Health Promotion Program
Number analyzed (Participants) | 6
percentage of glycosolated hemoglobin | -0.5 (0.5)

ADVERSE EVENTS:
Arm/Group | Health Promotion Program
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No